CLINICAL TRIAL: NCT03226483
Title: Intraoperative Radiotherapy After the Resection of Brain Metastases - a Phase II Feasibility Study
Brief Title: Intraoperative Radiotherapy After the Resection of Brain Metastases
Acronym: INTRAMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Stefanie Brehmer, MD, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-638N-MA
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Brain Metastases
Keywords: Brain Metastases; Intraoperative Radiotherapy; Neurosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative radiotherapy (Experimental): After neurosurgical resection and proven metastasis (frozen section) a local intraoperative radiotherapy with soft energy x-rays is applied to the resection cavity.
  To perform this an applicator is inserted into the situs in the tightest fit rule. The highest possible dose between 30-20 Gy is chosen depending on nearby risk structures (Optic nerve, brainstem) is prescribed. After radiotherapy the applicator is removed and the surgery will be finished in standard way.
  Interventions: Radiation: Intraoperative Radiotherapy

INTERVENTIONS:
Radiation: Intraoperative Radiotherapy — Intraoperative Radiotherapy is performed with a mobile radiation device emitting soft energy x-rays in a spherical way. Different size applicators are available to cover the resection cavity after the tightest fit rule.

SUMMARY:
INTRAMET examines prospectively the effectiveness of an intraoperative radiotherapy immediate after the surgical resection of brain metastases. Patients won't receive further radiation therapy of the intraoperatively treated lesion.

DETAILED DESCRIPTION:
Brain metastases occur in up to 40% of all patients diagnosed with systemic cancer. Without adjuvant radiotherapy after resection of space occupying lesions local recurrence rates are high. That is why guidelines recommend a cavity boosting with x-rays. External beam radiotherapy can lower the risk of local recurrence but means longer hospitalization, prolongs the time to systemic salvage therapies and bears risks of radionecrosis and leucoencephalopathy with neurological and cognitive decline. A solution for this problem could be onetime intraoperative radiotherapy (IORT) with soft x-rays to sterilize the resection cavity, which may provide both: freedom from local recurrence fast track salvage therapy initiation.

INTRAMET is a single institution, open-label, prospective, phase 2 feasibility study for intraoperative radiotherapy immediately following resection of brain metastases. 50 adult patients with resectable not dural brain metastases should be treated in surgery after tumor resection with IORT with 20-30Gy prescribed to the margin of the resection cavity. The highest dose tolerable to surrounding risk structures (N. opticus, brainstem) should be used.

With this method, the investigators hope to show similar local control rates to postoperative external beam radiotherapy in line with guideline recommendations with less patient hospitalization and faster start of rescue therapies which could lead to a favorable overall outcome and less cognitive side effects.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance index ≥ 50%
* MRI T1 Gadolinium enhancing non-dural resectable lesion
* Informed consent
* Adequate birth control
* Frozen section confirms metastasis
* Adequate distance to optic nerve and brainstem

Exclusion Criteria:

* Dural lesions or meningeal carcinomatosis
* Frozen section reveals glioma, lymphoma,small cell lung cancer or germinoma
* Psychiatric or social condition interfering compliance
* Contraindication against anesthesia, surgery, MRI and/or Gadolinium
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Median local progression-free-survival | 2 years
  Rate of recurrence of the treated lesion in the brain

SECONDARY OUTCOMES:
Overall-survival | 5 years
  Survival differentiated between death due to systemic cancer progress and death due to cerebral progress
Time to further therapy | 6 month
  Time to further cancer therapy (e.g. salvage chemotherapy)
Patients cognitive performance | 5 years
  Neuropsychological battery
Patients quality of life | 5 years
  Patient questionary
Global progression-free-survival | 2 years
  Systemic cancer progression-free-survival
Regional progression-free-survival | 2 years
  Progression-free survival concerning other brain metastases
Intraoperative radiotherapy caused dose-limiting toxicities | 6 month after intervention
  Occurrence of wound healing disorders or infection requiring surgical revision, cerebral bleeding or ischemia, radionecrosis requiring surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Brehmer, MD, Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Germany